CLINICAL TRIAL: NCT00061789
Title: SPECT Imaging of Alpha 4 Beta 2 Nicotinic Acetylcholine Receptors Using [(123)I]5-I-A-85380 in Schizophrenia
Brief Title: Imaging of Brain Receptors in Healthy Volunteers and in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030003; 03-M-0003
Record Dates: First submitted 2003-06-04; First posted 2003-06-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; SPECT; Nicotinic Acetylcholine Receptors; Cigarette Smoking; Cognitive Dysfunction; Reproducibility; Quantification; Healthy Volunteer; HV
MeSH Terms: conditions — Schizophrenia; Cigarette Smoking; Cognitive Dysfunction

INTERVENTIONS:
Drug: SPECT Imaging of Nicotinic Acetylcholine Receptors in Brain

SUMMARY:
This study will use single photon emission computed tomography (SPECT) to study brain nicotine receptors (proteins on the surface of brain cells) in healthy subjects and in patients with schizophrenia. Autopsy findings in patients with schizophrenia show changes in their nicotine receptors. This study will use SPECT to look at these receptors in living schizophrenia patients and compare them with those in healthy subjects.

The following individuals between 21 and 50 years of age (or between 21 and 80 years of age for Group 1 only) are eligible for this study: healthy non-smokers (Group 1); schizophrenia patients who smoke (Group 2); schizophrenia patients who do not smoke (Group 3); healthy smokers (Group 4); healthy non-smokers (Group 5). Patients with schizophrenia must be taking olanzapine (Zyprexa) or risperidone (Risperdal) for at least 6 months. All candidates will be screened at the first visit. Group 1 participants will have three more visits; Groups 2 through 5 will have two more visits.

Visit 1

All participants will be screened with physical and neurological examinations; blood and urine tests; and neuropsychological tests to assess their ability to learn and remember words and numbers, to pay attention, and to quickly perform motor tasks, such as putting pegs into a piece of wood. In addition, they will have an eye movement test and event-related potential testing. For the eye test, the subject sits in a chair and leans forward with the chin on a chin rest. A band is tied around the head and very small amounts of invisible (infrared) light are shined into the eyes. The light is reflected back and measured. Wire electrodes are placed around the area of the eye and cheek to monitor eye blinks and eye movements. Subjects are asked to follow a light with their eyes and to look away from a light. For event- related potential testing, electrodes are placed on the scalp, forehead and cheeks, and brain activity is recorded while the subject identifies particular pictures and sounds.

Visit 2 (and Visit 3 for Group 1)

Participants will have a SPECT scan. On the night before the scan, the day of the scan, and for 4 days after the scan, subject take an oral dose of potassium iodide to protect the thyroid gland from the radioactive tracer used in the SPECT procedure. (Individuals allergic to potassium iodide will take potassium perchlorate instead.) For the SPECT scan, small radioactive markers containing 99mTc are glued to the subject's head. Two catheters (thin, flexible tubes) are placed in veins in the arms to inject the radioactive tracer [123I]5-I-A-85380 and to draw blood samples. During the scan, the subject lies on a bed with his or her head held still with a headholder. The scans are taken over a 9-hour period after injection of the tracer injection. An electrocardiogram, respiration, and blood pressure measures are taken before injection of [123I]5-I-A-85380, then 5 minutes after the injection, and again 30 to 60 minutes after the injection. Breath samples are collected every 60 minutes. Blood and urine samples are collected 5 to 6 hours after starting the scan. Group 1 subjects will have a second SPECT scan within 4 weeks of the first.

Visit 3 (Visit 4 for Group 1)

Participants will have a magnetic resonance imaging (MRI) scan. For this procedure, the subject lies on a table that slides into a narrow metal cylinder with a strong magnetic field for the scan. The scanner uses a magnetic field and radio waves to produce images that show structural and chemical changes in tissues. The test lasts up to 1 hour.

DETAILED DESCRIPTION:
Abnormalities of nicotinic acetylcholine system in schizophrenia are implied by the high prevalence of cigarette smoking. Because animal and human studies have shown that nicotinic acetylcholine receptors (nAChRs) play an important role in cognitive function, cognitive deficits in schizophrenia also suggest abnormalities in these receptors. Postmortem studies showed abnormalities in high affinity nAChRs in these patients but the direction of the abnormalities (increase or decrease) were not consistent probably because it is difficult to control the effects of cigarette smoking and neuroleptics in such studies. In vivo imaging studies are necessary to study relationship between nAChRs and psychiatric symptoms including cognitive impairments.

We plan to use a new single photon emission computed tomography (SPECT) tracer, [(123)I]5-I-A-85380, which appears suitable for imaging the high affinity Alpha 4 Beta 2 subtype of nAChRs. We plan to compare four groups, 1) schizophrenia smokers, 2) schizophrenia non-smokers, 3) healthy smokers, and 4) healthy non-smokers. All patients will be on stable doses of olanzapine or risperidone. In addition to comparing [(123)I]5-I-A-85380 binding among these groups, relationship will be studied between psychiatric symptoms or cognitive dysfunction and the SPECT measurement of the receptors. Further, to study the reliability of the SPECT measurement, a test retest study will be preformed in healthy subjects with a wide range. The proposed study will explore the roles of nAChRs in the psychiatric symptoms, particularly the cognitive deficits in schizophrenia, which is the central impairment of this disorder. New findings in this research will lead to enhanced treatment of the cognitive deficits.

ELIGIBILITY:
INCLUSION CRITERIA:

Controls-Group 1:

Healthy Diagnosis;

21-80 years;

No Cigarette Smoking;

Plasma Cotinine less than 3 ng/mL;

No olanzapine or risperidone

Smoker Patients-Group 2:

Diagnosis of Schizophrenia;

21-50 years;

Cigarette Smoking greater than 20 per day and greater than 5 years;

Plasma Cotinine greater than 100 ng/mL;

Olanzapine or risperidone greater than 6 mo. and same dose for 2 weeks

Non-Smoker Patients-Group 3:

Diagnosis of Schizophrenia;

21-50 years;

No Cigarette Smoking;

Plasma Cotinine less than 3 ng/mL;

Olanzapine or risperidone greater than 6 mo. and same dose for 2 weeks

Smoker Controls-Group 4:

Healthy Diagnosis;

21-50 years;

Cigarette Smoking greater than 20 per day and greater than 5 years;

Plasma Cotinine greater than 100 ng/mL;

No olanzapine or risperidone

Non-Smoker Controls-Group 5:

Healthy Diagnosis;

21-50 years;

No Cigarette Smoking;

Plasma Cotinine less than 3 ng/mL;

No olanzapine or risperidone

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2003-02; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States